CLINICAL TRIAL: NCT06527989
Title: Prophylactic Antibiotic in Subtalar Fusion Surgery: 24 Hours Versus 5 Days
Brief Title: Prophylactic Antibiotic in Subtalar Fusion Surgery
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ibram romany labib nashed, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: antibiotic prophylaxis
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ceftriaxone

STUDY DESIGN:
Intervention Model Description: Preoperative: IV administration of prophylactic antibiotic 2gram ceftriaxone 30 to 60 min before surgical incision Intraoperative: if there is blood loss
  Postoperative:
  * Group A : Single dose 2grams of ceftriaxone in 1st 24 hr
  * Group B: Multiple doses 2 grams of ceftriaxone every 24 hrs for 5 days Follow up assessment of surgical wound 2 weeks after surgery for both groups then lately after 3 months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceftriaxone 2 grams (Experimental): Single dose 2grams of ceftriaxone in 1st 24 hr Postoperative
  Interventions: Drug: Ceftriaxone 2000 mg
- ceftriaxone 10 grams (Experimental): Multiple doses 2 grams of ceftriaxone every 24 hrs for 5 days
  Interventions: Drug: Ceftriaxone 2000 mg

INTERVENTIONS:
Drug: Ceftriaxone 2000 mg — antibiotic prophylaxis
  Other Names: ceftriaxone

SUMMARY:
Assessment of surgical site infection when using postoperative antibiotic prophylaxis in subtalar fusion surgery 24hours versus 5 days

DETAILED DESCRIPTION:
Infection in orthopedic surgery is one of the most dreaded complications. Antibiotic prophylaxis should be utilized routinely in foot and ankle surgeries involving bone, utilizing hardware and prosthetic joints.

It is appropriate for the antibiotics to be administered within 60 minutes prior to surgery, discontinued within 24 hours after surgery, given prior to tourniquet inflation, and utilized routinely in prolonged foot and ankle surgery cases.

Narrow spectrum antibiotics covering Staphylococcus aureus should be utilized for prophylaxis in patients without a history of resistant infection. According to American Society of Health System Pharmacists (ASHP) cefazolin was the most used antibiotic in preoperative prophylaxis, combination of cefazolin with gentamicin was the second common regimen while 3rd generation cephalosporin were 3rd widely used antibiotics.

The controversy persists in administration of antibiotics varying from a single dose to 3 doses to 5 days or 14 days. In subtropical country, with a hot and humid climate is a conducive environment for both Gram-positive and Gram-negative bacterial colonization of skin. Therefore, we need studies tailored to our environment in Egypt Prevention of SSIs is critical for the health of patients, Economic efficiency, Antibiotic resistance considerations In conclusion, in many ways, the topic of prophylactic antibiotics in elective foot and ankle surgery is an unusual one, in that a relative divide exists between empirical science and common practice.

ELIGIBILITY:
Inclusion Criteria:

1. posttraumatic subtallar osteoarthritis
2. adult age 18 up to 60
3. good skin condition healthy

Exclusion Criteria:

1. comorbidities such as Diabetes Mellitus, Autoimmune diseases
2. previous foot surgery
3. wounds near surgical incision
4. skin infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
assessment of incidence rate of surgical site infection | baseline
  surgical site infection are further classified as either superficial or deep. Superficial infections involve only the skin and subcutaneous tissue, whereas deep infections involve deep tissue spaces or organs

CONTACTS AND LOCATIONS:
Overall Officials: Wael Y Eladly, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dayton P, DeVries JG, Landsman A, Meyr A, Schweinberger M. American college of foot and ankle surgeons' clinical consensus statement: perioperative prophylactic antibiotic use in clean elective foot surgery. J Foot Ankle Surg. 2015 Mar-Apr;54(2):273-9. doi: 10.1053/j.jfas.2015.01.004. Epub 2015 Jan 24. PMID 25631195
- [Result] Dhammi IK, Ul Haq R, Kumar S. Prophylactic antibiotics in orthopedic surgery: Controversial issues in its use. Indian J Orthop. 2015 Jul-Aug;49(4):373-6. doi: 10.4103/0019-5413.159556. No abstract available. PMID 26229155
- [Result] Upadhyyaya GK, Tewari S. Enhancing Surgical Outcomes: A Critical Review of Antibiotic Prophylaxis in Orthopedic Surgery. Cureus. 2023 Oct 27;15(10):e47828. doi: 10.7759/cureus.47828. eCollection 2023 Oct. PMID 38022210